CLINICAL TRIAL: NCT01758835
Title: Evaluation of Different Non-operative Treatment Protocols of ER-stress Negative Weber-B Unimalleolar Ankle Fractures. A Prospective Randomized Multicenter Trial.
Brief Title: PRCT-study of Different Non-operative Treatment Protocols of ER-stress Negative Weber-B Unimalleolar Ankle Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Harri Pakarinen, Orthopedic surgeon, MD, PhD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OYSrctAnkle5
Record Dates: First submitted 2012-12-21; First posted 2013-01-01 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Lateral Malleolus Fractures
Keywords: ER-stress-test negative; unimalleolar; fibula; Weber-B fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Splints; POLR1G protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Splint 3 weeks (Active Comparator): Removable ankle brace/splint
  Interventions: Other: Splint 3 weeks
- Cast 3 weeks (Active Comparator): Below-the-knee cast (glass fiber)
  Interventions: Other: Cast 3 weeks
- Cast 6 weeks (Active Comparator): Below-the-knee cast (glass fiber)
  Interventions: Other: Cast 6 weeks

INTERVENTIONS:
Other: Splint 3 weeks — A removable orthosis/splint. Dynacast/Ortho-Glass AS (BSN Medical). Splint is used for 3 weeks and no additional support is used after splint removal.
  Arms: Splint 3 weeks
Other: Cast 3 weeks — A standard short boot cast from proximal tibia to MTP I-V joint line. Cast is made from 3M Scotchcast. Cast is removed after 3 weeks and no additional support is used after cast removal.
  Arms: Cast 3 weeks
Other: Cast 6 weeks — standard short boot cast from proximal tibia to MTP I-V joint line. Cast is made from 3M Scotchcast. Cast is changed after 3 weeks and removed after 6 weeks. No additional support is used after cast removal.
  Arms: Cast 6 weeks

SUMMARY:
PRCT multicenter study to evaluate non-operative treatment protocols for treating ER-stress negative unimalleolar Weber-B type fibular fractures. Groups are: 1. 3 weeks in a removable splint 2. 3 weeks in a cast and 3. 6 weeks in a cast. Follow-up visits at 3, 6 and 12 weeks and after 1 and 2 years after injury. In each time X-rays laterally and mortise projections. Ankle functional outcome questionnaires: Olerud-Molander score, FAOS RAND-36 and VAS in follow up-visits 6 and 12 weeks and 1 and 2 year.

DETAILED DESCRIPTION:
Prospective randomized controlled multicenter study to evaluate non-operative treatment protocols for treating ER-stress negative unimalleolar Weber-B type fibular fractures. Groups are: 1. 3 weeks in a removable splint 2. 3 weeks in a cast and 3. 6 weeks in a cast. Follow-up visits at 3, 6 and 12 weeks and after 1 and 2 years after injury. In each time X-rays laterally and mortise projections. Ankle functional outcome questionnaires: Olerud-Molander score, FAOS RAND-36 and VAS in follow up-visits 6 and 12 weeks and 1 and 2 year.

ELIGIBILITY:
Inclusion Criteria:

* Stable Weber-B type fibula fracture
* ER-stress negative
* 16 or over years old
* Willingness to participate on study proved by a signature and date
* Walking without aid before accident
* Treatment started within 7 days from injury

Exclusion Criteria:

* Prior ankle fracture or significant fracture in the area of ankle or leg
* Bilateral ankle fracture
* Pathological fracture
* Diabetes mellitus or an other significant periferial neuropathy
* municipality of Residence in some else catchment area than Oulu university hospital or Tampere university hospital
* Patient's understanding or co-operation inadequate

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Olerud-Molander score | 1 year
  Ankle functional outcome measure

SECONDARY OUTCOMES:
FAOS | 1 year
  Foot and Ankle Outcome Score
VAS | 1 year
  Visual Analogue Scale pain and function
RAND 36 Health item survey | 1 year
  Quality of life measurement
Fracture healing | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Harri J Pakarinen, MD, PhD, Study Director — Oulu University Hospital; Tero HJ Kortekangas, MD, Principal Investigator — Oulu University Hospital
Locations (1):
- OYS, kirurgian klinkka, Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kortekangas T, Haapasalo H, Flinkkila T, Ohtonen P, Nortunen S, Laine HJ, Jarvinen TL, Pakarinen H. Three week versus six week immobilisation for stable Weber B type ankle fractures: randomised, multicentre, non-inferiority clinical trial. BMJ. 2019 Jan 23;364:k5432. doi: 10.1136/bmj.k5432. PMID 30674451